CLINICAL TRIAL: NCT00944099
Title: Eating Frequency Prescription for a Behavioral Weigh Loss Intervention
Brief Title: Lifestyle, Eating, and Activity Patterns
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHA 09PRE2020150
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obesity
Keywords: intervention studies; feeding behavior; eating frequency; weight loss; dietary intake
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazing (Experimental): participants will be given an eating frequency prescription to eat every 2 to 3 hours
  Interventions: Behavioral: Behavioral weight loss intervention
- Three Meals (Experimental): participants will be given an eating frequency prescription of eating 3 meals per day
  Interventions: Behavioral: Behavioral weight loss intervention

INTERVENTIONS:
Behavioral: Behavioral weight loss intervention — both conditions will receive an identical dietary prescription, low-calorie and less than 30% calories from fat and an identical physical activity goal of 200 minutes of moderate-intense physical activity per week during a 6 month behavioral weight loss program

SUMMARY:
The purpose of this research is to test the effect of manipulating eating frequency on hunger and the reinforcing value of food in 50 overweight/obese adults participating in a 6-month behavioral weight loss intervention.

DETAILED DESCRIPTION:
Previous observational and experimental research suggests that increased eating frequency is related to lower weight, body mass index (BMI)and body fatness. It is proposed that eating frequently during the day reduces overall energy consumed by preventing the development of excessive hunger. As elevated hunger increases the reinforcing value of food, and greater intake occurs when the reinforcing value of food increases, eating frequently during the day may be a dietary strategy that can aid with reducing energy intake and improving weight loss during a behavioral weight control program. Therefore, the purpose of this proposed research is to test the effect of manipulating eating frequency on hunger and the reinforcing value of food in 50 overweight/obese adults participating in a 6-month behavioral weight loss intervention. Participants will be randomized to 1 of 2 conditions: 1) a condition in which participants will be given an eating frequency prescription to eat every 2 to 3 hours (Grazing); or 2) a condition in which participants will be given an eating frequency prescription of eating 3 meals per day (Three Meals). Both conditions will receive an identical dietary prescription, a low-calorie (1200 to 1500 kcals/d), low-fat (≤ 30% kcals from fat) diet and an identical physical activity goal of 200 minutes of moderate-intense physical activity per week. Additionally, both conditions will receive an identical state-of-the-art, 6-month, behavioral weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 27 and 45 kg/m2

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* report being unable to walk 1/4 mile without stopping
* report major psychological disease or organic brain syndromes
* report a diagnosis of type I or type II diabetes
* are currently participating in a weight loss program, are taking weight loss medication, have had surgery for weight loss, or have lost > 5% of their body weight in the past 6 months
* are currently participating in a program that manipulates their eating habits
* intent to move outside of the East Tennessee area within the time frame of the intervention
* are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the intervention
* are unwilling to attend group intervention meetings, assessments, or complete a food diary for the duration of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
eating occasions per day | 0, 3, and 6 months
hunger and reinforcing value of food | 0, 3, and 6 months

SECONDARY OUTCOMES:
energy and percent calories from fat intake | 0, 3, and 6 months
body weight, percent body fat, percent fat free mass | 0, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Bachman, MS, MPH, RD, Principal Investigator — University of Tennessee; Hollie A Raynor, PhD, RD, Study Chair — University of Tennessee
Locations (1):
- Healthy Eating and Acitivty Laboratory, University of Tennessee, Knoxville, Tennessee, United States